CLINICAL TRIAL: NCT00886860
Title: The Comparison of Efficacy for Cervical Ripening in Labor Induction Between Titrated and Conventional Oral Misoprostol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Kusol Russameecharoen, MD., Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 091/2552(EC2)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Cervical Ripening; Labor Induction
Keywords: Efficacy; Cervical ripening/Labor induction; Titrated oral misoprostol/Conventional oral misoprostol; Term pregnancy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional oral misoprostol (Active Comparator): misoprostol 50 micrograms oral every 4 hours until cervical dilatation 3 centimeters
  Interventions: Drug: misoprostol
- titrated oral misoprostol (Experimental): misoprostol 20 micrograms oral every hour until cervical dilatation 3 centimeters
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — misoprostol 50 micrograms oral every 4 hours until cervical dilatation 3 cm
  Other Names: cytotec
  Arms: conventional oral misoprostol
Drug: misoprostol — misoprostol 20 micrograms oral every hours until cervical dilatation 3 cm
  Other Names: cytotec
  Arms: titrated oral misoprostol

SUMMARY:
The purpose of this study is to compare the efficacy for cervical ripening in labor induction between titrated and conventional oral misoprostol

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old or more
* singleton pregnancy at 37 weeks gestation or more
* cephalic presentation
* reassuring fetal heart rate pattern
* admission for labor induction due to medical or obstetrical conditions
* bishop score less than 6
* giving consent and having signed the consent form for this study

Exclusion Criteria:

* parity more than 3
* estimated fetal weight more than 3,500 grams
* non-reassuring fetal heart rate pattern
* having contraindication for vaginal delivery
* previous uterine scar
* suspected abruptio placenta with non-reassuring fetal heart rate pattern
* abnormal bleeding per vagina, except bloody show
* PROM
* having underlying cardiac, hepatic, or renal diseases
* having history of allergy to misoprostol or prostaglandin analogues
* cervical dilatation 3 centimeters or more
* uterine contraction 3 times or more in 10 minute

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
success rate of cervical ripening in labor induction | 12 hours after intervention

SECONDARY OUTCOMES:
number of vaginal delivery | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kusol Russameecharoen, MD, Study Director — Siriraj Hospital, Mahidol University Bangkok, Bangkok, Thailand
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Thaisomboon A, Russameecharoen K, Wanitpongpan P, Phattanachindakun B, Changnoi A. Comparison of the efficacy and safety of titrated oral misoprostol and a conventional oral regimen for cervical ripening and labor induction. Int J Gynaecol Obstet. 2012 Jan;116(1):13-6. doi: 10.1016/j.ijgo.2011.07.027. Epub 2011 Sep 28. PMID 21959071